CLINICAL TRIAL: NCT07280975
Title: Comparative Outcomes of Polyglactin Versus Polypropylene Sutures for Rectus Sheath Closure: A Randomized Controlled Trial
Brief Title: Comparing Polyglactin vs Polypropylene Sutures for Rectus Sheath Closure
Acronym: PolySuture
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Reading Hospital, Pakistan (Other Government)
Responsible Party: Principal Investigator, Dr. Waseem Ullah, Registrar, General Surgery, Lady Reading Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 563/LRH/MTI
Record Dates: First submitted 2025-11-28; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain; Wound Dehiscence; Surgical Site Infection (SSI); Incisional Hernia; Rectus Sheath Closure; Abdominal Surgery
Keywords: Polyglactin Sutures; Polypropylene Sutures; Non-Absorbable Sutures; Postoperative Complications; Midline Laparotomy
MeSH Terms: conditions — Chronic Pain; Surgical Wound Infection; Incisional Hernia; Postoperative Complications | interventions — Polyglactin 910; Sutures; Polypropylenes

STUDY DESIGN:
Intervention Model Description: This is a parallel-group design, where participants are assigned to one of two treatment arms (polyglactin or polypropylene). Both arms will undergo the same procedure but with different suture materials for rectus sheath closure.
Who Masked: Participant, Outcomes Assessor
Masking Description: This study is single-blind, meaning the participants do not know which suture material they received. The outcomes assessor (surgeon) will also be blinded to the group allocation to reduce bias in outcome assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polyglactin 910 (Vicryl) Suture for Rectus Sheath Closure (Experimental): In this arm, participants will undergo rectus sheath closure using polyglactin 910 (Vicryl), a synthetic absorbable braided suture. This material is designed to provide temporary wound support during the healing process, with predictable hydrolytic degradation over 56-70 days. The intervention involves continuous suturing of the rectus sheath, with the suture size being 1 (USP). The primary aim is to evaluate postoperative outcomes such as incisional hernia, surgical site infections, wound dehiscence, and chronic pain, using polyglactin sutures for abdominal wall closure.Polyglactin 910 (Vicryl) Suture for Rectus Sheath Closure
  Interventions: Procedure: Polyglactin 910 (Vicryl) Suture
- Polypropylene (Prolene) Suture for Rectus Sheath Closure (Active Comparator): In this arm, participants will undergo rectus sheath closure using polypropylene (Prolene), a non-absorbable monofilament suture. Polypropylene is known for its high tensile strength and biocompatibility, providing long-term mechanical support without being absorbed by the body. The intervention will involve continuous suturing of the rectus sheath, using a size 1 (USP) suture. The main focus will be to assess the incidence of complications such as incisional hernia, surgical site infection, wound dehiscence, and chronic pain following closure with polypropylene sutures.
  Interventions: Procedure: Polypropylene (Prolene) Suture

INTERVENTIONS:
Procedure: Polyglactin 910 (Vicryl) Suture — Polyglactin 910 (Vicryl) is an absorbable synthetic multifilament suture material used for rectus sheath closure following laparotomy. This suture material undergoes hydrolytic degradation over a period of 56-70 days and retains approximately 75% of its tensile strength at 2 weeks and 50% at 3 weeks, which aligns with the typical biological timeline for fascial healing. It is used to approximate the anterior rectus sheath with a continuous suturing technique.
  Arms: Polyglactin 910 (Vicryl) Suture for Rectus Sheath Closure
Procedure: Polypropylene (Prolene) Suture — Polypropylene (Prolene) is a non-absorbable monofilament suture material used for rectus sheath closure following laparotomy. It provides long-term mechanical support for abdominal wall closure and does not degrade over time. The suture material maintains its tensile strength indefinitely and is known for its high biocompatibility, minimal tissue reaction, and resistance to infection due to its monofilament structure. It is applied using a continuous suturing technique.
  Arms: Polypropylene (Prolene) Suture for Rectus Sheath Closure

SUMMARY:
This randomized controlled trial aims to compare the outcomes of Polyglactin (Vicryl) versus Polypropylene (Prolene) sutures for rectus sheath closure in patients undergoing midline laparotomy. The study will evaluate the rates of incisional hernia, surgical site infection (SSI), wound dehiscence, chronic pain, and suture sinus formation. Participants aged 18-70 years, undergoing either elective or emergency laparotomy, will be randomly assigned to receive either Polyglactin or Polypropylene sutures. The primary outcome measure is the incidence of incisional hernia at 6 months, with secondary outcomes including SSI, wound complications, and chronic pain. The study is particularly important in the context of Pakistan, where such comparative data is limited, and aims to provide evidence-based recommendations for optimal suture material selection in general surgery.

DETAILED DESCRIPTION:
Study Design This randomized controlled trial is designed to compare the outcomes of two suture materials-Polyglactin 910 (Vicryl) and Polypropylene (Prolene)-for rectus sheath closure after midline laparotomy. The study will be conducted at the Department of General Surgery, Lady Reading Hospital, Peshawar, over 12 months. Participants will be randomly assigned to two groups: Group A (Polyglactin) and Group B (Polypropylene). The primary outcome is the rate of incisional hernia at 6 months postoperatively. Secondary outcomes include surgical site infection (SSI), wound dehiscence, chronic pain, and suture sinus formation.

■ Participants The study will include patients aged 18 to 70 years undergoing elective or emergency midline laparotomy with clean or clean-contaminated wounds (CDC Class I or II).

Inclusion Criteria:

Aged 18-70 years

Elective or emergency laparotomy

Clean or clean-contaminated wounds

Ability to provide informed consent

Availability for 6-month follow-up

Exclusion Criteria:

Contaminated or dirty wounds (CDC Class III or IV)

Immunocompromised patients (e.g., on steroids, chemotherapy, HIV)

Prior midline laparotomy with incisional hernia

Severe malnutrition (BMI <16 kg/m² or albumin <2.5 g/dL)

Pregnancy

Requirement for temporary abdominal closure or planned reoperation

■ Interventions

Polyglactin (Vicryl): A synthetic absorbable braided suture composed of glycolide and lactide copolymers. It is absorbed by hydrolysis over 56-70 days, providing temporary wound support during healing.

Polypropylene (Prolene): A synthetic non-absorbable monofilament suture known for its permanent tensile strength and excellent biocompatibility, offering long-term mechanical support and minimal tissue reaction.

Outcome Measures

Primary Outcome:

Incidence of incisional hernia at 6 months, confirmed by clinical examination and ultrasound if necessary.

Secondary Outcomes:

Surgical Site Infection (SSI): Defined as an infection occurring within 30 days post-surgery, classified as superficial, deep, or organ/space.

Wound Dehiscence: Partial or complete disruption of the abdominal wall closure within 30 days post-surgery.

Chronic Pain: Persistent pain at the surgical site lasting more than 3 months, assessed using the Visual Analog Scale (VAS).

Suture Sinus Formation: Chronic draining tract related to the suture material.

Statistical Analysis Data will be analyzed using SPSS version 26. Chi-square tests will compare proportions of complications between the two groups, and relative risk will be calculated with 95% confidence intervals. Stratified analysis will assess the impact of potential modifiers such as age, gender, and comorbidities (e.g., diabetes, hypertension).

Potential Impact The findings from this study aim to improve surgical outcomes in Pakistan and similar settings. By identifying the more effective suture material for rectus sheath closure, this research will help guide clinical practices, reducing common complications like incisional hernia and infection. It may also contribute to better surgical standards in regions lacking high-quality comparative data.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years.
2. Type of Surgery: Patients undergoing elective or emergency midline laparotomy.
3. Wound Classification: Clean or clean-contaminated wounds (CDC Class I or II).
4. Ability to Provide Informed Consent: Participants must be able to understand and sign the informed consent form.
5. Availability for Follow-Up: Participants must be available for 6 months follow-up.

Exclusion Criteria:

1. Contaminated or Dirty Wounds: Patients with CDC Class III or IV wounds.
2. Immunocompromised Conditions: Patients on steroids, chemotherapy, or those with HIV.
3. Previous Midline Laparotomy with Incisional Hernia: Patients who have a history of incisional hernia after midline laparotomy.
4. Severe Malnutrition: Patients with BMI < 16 kg/m² or albumin < 2.5 g/dL.
5. Emergency Laparotomy with Hemodynamic Instability: Patients who are unstable or in a critical condition.
6. Pregnancy: Pregnant women.
7. Need for Temporary Abdominal Closure or Planned Reoperation: Patients requiring staged reoperation or temporary closure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Incisional Hernia rate | 6 months postoperatively
  The primary outcome will assess the rate of incisional hernia at 6 months post-surgery in patients who undergo rectus sheath closure with either Polyglactin 910 (Vicryl) or Polypropylene (Prolene) sutures.

SECONDARY OUTCOMES:
Surgical Site Infection (SSI) Rate | 30 days post-surgery
  This outcome will measure the occurrence of any surgical site infection (SSI) within 30 days postoperatively.
Suture Sinus Formation | 6 months post-surgery
  The occurrence of chronic draining tracts at the incision site, which are associated with the suture material.
Chronic Pain (Visual Analog Scale, VAS ≥4) | 3 months post-surgery
  The presence of chronic pain at the surgical site lasting more than 3 months postoperatively, assessed using the Visual Analog Scale (VAS), where the VAS is a 10-point scale ranging from 0 (no pain) to 10 (worst possible pain). A score of 4 or higher indicates the presence of clinically significant chronic pain.
Wound Dehiscence | 30 days post-surgery
  The occurrence of wound dehiscence, defined as partial or complete disruption of the rectus sheath, within 30 days post-surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Lady Reading Hospital, Department of General Surgery, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) that will be shared includes de-identified demographic information, surgical details, treatment outcomes, and relevant follow-up data (e.g., wound healing, incidence of complications, pain scores, and hernia occurrence). This will provide valuable insight into the comparative efficacy of polyglactin versus polypropylene sutures for rectus sheath closure. The data will be available to qualified researchers after the primary results have been published and the study is concluded.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The IPD and supporting information will be accessible to qualified researchers affiliated with academic, medical, or research institutions who are involved in the study of similar surgical outcomes or suture materials. These researchers will be able to access:
  De-identified patient data (demographic, clinical outcomes, complications) Study protocol, SAP, ICF, CSR, and analytic code
Access Criteria: Access will be granted through a secure online platform (such as a data repository) after a formal request and approval by the institution's data access committee. Researchers will be required to adhere to confidentiality agreements and data protection regulations.